CLINICAL TRIAL: NCT03563508
Title: A Cone-beam Computed Tomography Study of Root and Root Canal Morphology of Maxillary Premolars in an Egyptian Subpopulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maysa mostafa Ahmed, Principal Investigator, Cairo University
Other Study IDs: cebd-cu-2018-05-31
Record Dates: First submitted 2018-05-30; First posted 2018-06-20 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-05

CONDITIONS: Morphology of Maxillary Premolars in Egyptian Subpopulation
Keywords: cone beam computed tomography; maxillary premolars; root canal anatomy; root canal morphology; Egyptian population

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBCT of Egyptian subpopulation: Cone-beam computed tomography (CBCT) of a sample of Egyptian subpopulation containing maxillary premolars for image assessment.

SUMMARY:
to date there is no detailed examination of the root and root canal system of maxillary first and second premolars in an Egyptian subpopulation. in this study the investigators do an Observational analysis of available records of cone-beam computed tomography (CBCT) of root and canal morphology in the permanent maxillary first and second premolars in this population

DETAILED DESCRIPTION:
Failure of endodontic treatment of upper first and second premolar because of presence of missed canals with lack of data of its morphological variations in the Egyptian population.There are different methods to study canal morphology as tooth clearing and root canal staining, conventional and digital radiographs, radiographic assessment enhanced with contrast media. Recently cone-beam computed tomographic (CBCT) images have been found to be useful in providing accurate anatomic details in 3 dimensions for diagnosis and treatment planning before endodontic therapy.

in this study the investigators do an Observational analysis of available records of cone-beam computed tomography (CBCT) of root and canal morphology in the permanent maxillary first and second premolars in this population

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans with minimum of one premolar.
* Maxillary premolars with fully formed apices

Exclusion Criteria:

* CBCT scans with all maxillary premolars missed.
* Maxillary premolars with open apices
* Maxillary premolars with root resorption
* Maxillary premolars with calcifications or extensive coronal restoration.
* Maxillary premolars with root canal fillings, posts, crown restorations.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: • CBCT of a sample of Egyptian subpopulation in Cairo governorate
Sampling Method: Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
root numbers in maxillary first and second premolars | year
  root

SECONDARY OUTCOMES:
Number of canals per root | year
  root canal
Type of root canal | year
  Categorical data

CONTACTS AND LOCATIONS:
Locations (1):
- CairoU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
A Cone-beam computed tomography study of root and root canal morphology of maxillary premolars in an Egyptian subpopulation

REFERENCES:
- [Background] Abella F, Teixido LM, Patel S, Sosa F, Duran-Sindreu F, Roig M. Cone-beam Computed Tomography Analysis of the Root Canal Morphology of Maxillary First and Second Premolars in a Spanish Population. J Endod. 2015 Aug;41(8):1241-7. doi: 10.1016/j.joen.2015.03.026. Epub 2015 May 5. PMID 25956606
- [Background] Celikten B, Orhan K, Aksoy U, Tufenkci P, Kalender A, Basmaci F, Dabaj P. Cone-beam CT evaluation of root canal morphology of maxillary and mandibular premolars in a Turkish Cypriot population. BDJ Open. 2016 Jan 29;2:15006. doi: 10.1038/bdjopen.2015.6. eCollection 2016. PMID 29607060
- [Background] Tian YY, Guo B, Zhang R, Yu X, Wang H, Hu T, Dummer PM. Root and canal morphology of maxillary first premolars in a Chinese subpopulation evaluated using cone-beam computed tomography. Int Endod J. 2012 Nov;45(11):996-1003. doi: 10.1111/j.1365-2591.2012.02059.x. Epub 2012 May 2. PMID 22551454